CLINICAL TRIAL: NCT03380962
Title: A Phase I/II Trial to Evaluate the Safety and Tolerability of Clazakizumab (Anti-IL-6 Monoclonal) to Eliminate Donor Specific HLA Antibodies (DSAs) and Improve Transplant Rates in Highly-HLA Sensitized Patients Awaiting Renal Transplant
Brief Title: Clazakizumab in Highly-HLA Sensitized Patients Awaiting Renal Transplant
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanley Jordan, MD (Other)
Responsible Party: Sponsor-Investigator, Stanley Jordan, MD, Director of the Kidney Transplant Program, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 48478
Record Dates: First submitted 2017-10-30; First posted 2017-12-21 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Kidney Failure, Chronic; End-Stage Renal Disease; Transplant Glomerulopathy; Transplant;Failure,Kidney; Kidney Transplant Failure and Rejection; Antibody-mediated Rejection; Kidney Transplant; Complications
Keywords: Donor-Specific Anti-HLA Antibodies; Kidney Transplantation; Donor Specific Antibody
MeSH Terms: conditions — Kidney Failure, Chronic; Rejection, Psychology | interventions — clazakizumab

STUDY DESIGN:
Intervention Model Description: Twenty enrolled study patients will receive study medication Clazakizumab (Vitaeris Inc; Vancouver Canada, BC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clazakizumab (Experimental): All twenty patients will receive clazakizumab monthly. Patients will receive up to 6 doses pre-transplantation. If patients are transplanted during the study, they will then receive 6 doses of clazakizumab (monthly) and a 6 month protocol biopsy will be performed. Based on the biopsy results and clinical labs PI will determine if patients should continue monthly doses for up to another 6 doses and day 330 post-transplantation. Patients who received 12 post-transplant doses of clazakizumab will then undergo a 12 month protocol biopsy.
  Interventions: Drug: Clazakizumab

INTERVENTIONS:
Drug: Clazakizumab — All patients will receive clazakizumab 25 mg subcutaneous injections (monthly) for a maximum of 18 injections.
  Other Names: Anti-IL-6 monoclonal

SUMMARY:
Patients who have had a previous allograft failure represent a major problem for transplant centers as they are highly-human leukocyte antigen (HLA) sensitized and unlikely to receive another transplant without significant desensitization. This single center, phase I/II, open label single-arm exploratory study focuses on enrolling twenty patients (ages 15-75) who will begin desensitization therapy to achieve HLA incompatible (HLAi) renal transplantation. Patients who qualify will receive up to 6 doses of clazakizumab 25 mg monthly pre-transplantation. If patients receive an HLAi transplant during the study, the participants will continue to receive another 6 monthly doses of clazakizumab 25 mg, followed by a 6 month protocol biopsy. Patients will continue another 6 doses over 6 months if improvements are seen after the 6th dose of clazakizumab. Patients who develop evidence of persistent allograft dysfunction may have non-protocol biopsies for cause. Patients who receive 12 doses of clazakizumab post-transplant will receive a 12M protocol biopsy.

DETAILED DESCRIPTION:
This is a single center, Phase I/II, open label single-arm exploratory study. The trial will primarily examine the safety and tolerability of clazakizumab given after consented and eligible patients begin desensitization therapy to achieve HLAi renal transplantation at Cedars-Sinai Medical Center. 20 subjects (ages 15 to 75) who are highly-HLA sensitized (HS) as determined by the cPRA ≥50% and are eligible for desensitization will be evaluated. All patients will be accrued from the renal transplant program at Cedars-Sinai Medical Center. Once desensitization begins, anti-HLA antibodies will be assessed which are associated with ABMR and/or graft loss. HLA antibodies will be detected using solid phase assay systems currently utilized at the Cedars-Sinai Medical Center HLA Laboratory. These anti-HLA antibodies may result naturally or from previous pregnancy, transfusions, or prior transplants. Patients treated with clazakizumab x 6 doses for desensitization will have blood sampling for HLA antibodies, and other monitoring blood samples as well as immunologic studies as outlined. If patients receive an HLAi transplant during the study, participants will receive the standard post-transplant immunosuppressive protocol, and clazakizumab 25 mg SC Q4W X 6 doses with immune monitoring as indicated.

Immune monitoring in blood samples for Treg, Tfh, Th17 and B-cell subsets as well as IL-6 and CRP monitoring will be carried out at the Cedars-Sinai Transplant Immunology Laboratory.

Patients identified as study participants will be HS and listed for HLAi renal transplantation at Cedars-Sinai Medical Center. Cedars-Sinai is a major U.S. desensitization center and performs ~80 HLAi renal transplants per-year. ~ 100 new HS patients are referred to Cedars-Sinai each year as potential candidates for desensitization. Eligible patients entering the study will initially receive PLEX (5-7 sessions) + IVIG and receive clazakizumab 25 mg SC one week post-IVIG. If no safety/tolerability/efficacy issues are observed after the initial dose, patients will receive 5 additional injections Q4W. If patients receive an HLAi transplant, clazakizumab will be continued for 6M post- transplant at 25mg SC Q4W for 6 doses (starting at Day 5 post-transplant). A protocol biopsy will be performed at 6M post-transplant to assess the allograft for evidence of ABMR, including C4d staining and TG using Banff 2015 criteria. Patients will continue another 6 doses over 6 months if improvements are seen after the 6th dose of clazakizumab. Patients who develop evidence of persistent allograft dysfunction may have non-protocol biopsies for cause. Patients who receive 12 doses of clazakizumab post-transplant will receive a 12M protocol biopsy. In the event a patient does not show improvement after receiving 6 doses of clazakizumab, no further treatment will be given and the patient will return at Day 365 for a final study visit. All subjects will be evaluated on an intent-to-treat basis. The subject accrual rate will be limited to no more than 1-2 subjects per month in the initial three months to assure safety to all subjects. Repeat laboratories will be performed at the completion of clazakizumab therapy to determine effect on levels and correlation with any potential events.

The subjects will be followed to determine if the use of clazakizumab for desensitization in this high risk transplant population is safe and without infectious risks. In addition, the investigators will determine the effects of clazakizumab treatment on HLA antibodies in efforts to improve access to HLAi transplants for these individuals. The investigators have previously reported acceptance criteria for HLAi kidney transplants. Renal biopsy assessments will be performed at 6M (per protocol) and 12M (for those who received 12 doses of therapy). The investigators will assess the transplanted patients to determine the number who sustain a viable and functioning kidney allograft as well. All subjects will be evaluated on an intent-to-treat basis. The subject accrual rate will be limited to no more than 1-2 subjects per month in the initial three months to assure safety to all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-75 years at the time of screening.
2. HS patients (cPRA≥50%) awaiting DD or LD kidney transplant on the UNOS list.
3. Previous history of pregnancies, blood transfusion and/or renal transplant.
4. Subject/Parent/Guardian must be willing to participate fully with study requirements.
5. Subject/Parent/Guardian must be able to understand and provide informed consent.
6. Pneumococcal vaccinated
7. Negative Tuberculin (ppd) placement result or negative Quantiferon TB gold results

Exclusion Criteria:

1. Multi-organ transplant (e.g. kidney and pancreas)
2. Intolerability to clazakizumab or other IL-6 inhibitor therapies
3. Lactating or pregnant females.
4. Women of child-bearing age and male partners of women of child-bearing age who are not willing or able to practice FDA-approved forms of contraception during study and for 5 months after last dose.
5. HIV-positive subjects.
6. Subjects who test positive for HBV by HBVeAg/DNA or HCV infection [positive Anti-HCV (EIA) and confirmatory HCV RIBA].
7. Subjects with latent or active TB. Subjects must have negative Quantiferon TB gold test result.
8. Recent recipients of any licensed or investigational live attenuated vaccine(s) within two months of the screening visit
9. A significantly abnormal general serum screening lab result defined as a ANC <2000, platelet count < 100 X 103/ml, an SGOT or SGPT > 1.5X upper limit normal.
10. Individuals deemed unable to comply with the protocol.
11. Subjects with active CMV or EBV infection as defined by CMV-specific serology (IgG or IgM) and confirmed by quantitative PCR with or without a compatible illness.
12. Use of investigational agents within 4 weeks of participation.
13. History or active Inflammatory Bowel Disease or Diverticular Disease or gastrointestinal perforation
14. Recent infection (within past 6 weeks of screening) requiring any antibiotic use (oral, parenteral or topical).
15. Present or previous (within 5 years) malignancy except for basal cell carcinoma, fully excised squamous cell carcinoma of the skin or non-recurrent (within 5 years) cervical carcinoma-in-situ

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in donor specific antibodies | Up to 21 months
  Assessment of HLA antibodies from baseline based on luminex assessments at multiple time points
Incidence of treatment related adverse effects of clazakizumab therapy | Up to 21 months
  Assessments of any side effects associated with clazakizumab administration and risk for infectious complications associated with clazakizumab therapy for desensitization of HS patients awaiting renal HLAi transplantation

SECONDARY OUTCOMES:
Change in Serum Creatinine | Up to 21 months
  Assessment of renal function by collecting Serum Creatinine (md/dl) at multiple time points
Incidence of ABMR episodes | Up to 12 months post-transplant
  Assessment of protocol biopsy results

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Jordan, MD, Principal Investigator — Cedars-Sinai Medical Center Comprehensive Transplant Center
Locations (1):
- Norko Ammerman, Los Angeles, California, United States

REFERENCES:
- [Background] Choi J, Aubert O, Vo A, Loupy A, Haas M, Puliyanda D, Kim I, Louie S, Kang A, Peng A, Kahwaji J, Reinsmoen N, Toyoda M, Jordan SC. Assessment of Tocilizumab (Anti-Interleukin-6 Receptor Monoclonal) as a Potential Treatment for Chronic Antibody-Mediated Rejection and Transplant Glomerulopathy in HLA-Sensitized Renal Allograft Recipients. Am J Transplant. 2017 Sep;17(9):2381-2389. doi: 10.1111/ajt.14228. Epub 2017 Mar 10. PMID 28199785
- [Derived] Fernando SC, Polkinghorne KR, Lim WH, Mulley WR. Early Versus Late Acute AMR in Kidney Transplant Recipients-A Comparison of Treatment Approaches and Outcomes From the ANZDATA Registry. Transplantation. 2023 Nov 1;107(11):2424-2432. doi: 10.1097/TP.0000000000004700. Epub 2023 Jun 16. PMID 37322595